CLINICAL TRIAL: NCT05448638
Title: Quality of Recovery Scores in Transversus Thoracic Muscle Plane Combined With Pectoral Nerves Block Versus Pectoral Nerves Block for Breast Cancer Surgery: a Randomized Controlled Trial
Brief Title: Transversus Thoracic Muscle Plane Combined With Pectoral Nerves Block for Breast Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Huifang Jiang, Principal Investigator, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-2022-348
Record Dates: First submitted 2022-07-03; First posted 2022-07-07 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transversus thoracic muscle plane block+pectoral nerves block (Experimental): the combination of transversus thoracic muscle plane and pectoral nerves blocks
  Interventions: Procedure: the combination of transversus thoracic muscle plane and pectoral nerves blocks
- pectoral nerves block (Active Comparator): the pectoral nerves block only
  Interventions: Procedure: the pectoral nerves block only

INTERVENTIONS:
Procedure: the combination of transversus thoracic muscle plane and pectoral nerves blocks — For the pectoral nerves block, 0.375% ropivacaine , 10ml was injected between the pectoralis major and pectoralis minor and 20 ml above the serratus anterior muscle. For the transversus thoracic muscle plane block, ropivacaine 0.375%,15ml was injected between the transversus thoracic muscle and the internal intercostal muscle.
  Arms: transversus thoracic muscle plane block+pectoral nerves block
Procedure: the pectoral nerves block only — For the pectoral nerves block, 0.375% ropivacaine , 10ml was injected between the pectoralis major and pectoralis minor and 20 ml above the serratus anterior muscle.
  Arms: pectoral nerves block

SUMMARY:
This is a prospective, randomized, controlled trial for evaluating the efficacy of addition of transversus thoracic muscle plane block to pectoral nerves block versus pectoral nerves block for quality of recovery scores in breast cancer surgery.

DETAILED DESCRIPTION:
The pectoral nerves (PECS) block cannot block the most internal mammary region, whereas a transversus thoracic muscle plane (TTP) block can. The combination of PECS and TTP blocks may be suitable for breast cancer surgery. We studied patients undergoing breast cancer surgery to assess whether the combination of PECS and TTP blocks provides better postoperative recovery than PECS block alone.

ELIGIBILITY:
Inclusion Criteria:

* female, 18-80 years of age
* American Society of Anesthesiologists physical status I-III
* patients having elective unilateral breast cancer surgery

Exclusion Criteria:

* contraindication to nerve block
* inability to understand or communicate with research personnel
* chronic use of opioids or nonsteroidal anti-inflammatory drugs
* pregnancy

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-08-05 (Actual)

PRIMARY OUTCOMES:
the quality of recovery-15 questionnaire (QoR-15) | at 24 hours after surgery
  The QoR-15 is a validated short-form postoperative quality of recovery score. Fifteen questions assess five domains of patient health-related quality of life: pain; comfort; physical independence; psychological support; and emotional state. Each question uses an 11-point rating scale, in which the maximum score is 150, denoting excellent recovery.
  1. Able to breathe easily
  2. Been able to enjoy food
  3. Feeling rested
  4. Have had a good sleep
  5. Able to look after personal toilet and hygiene unaided
  6. Able to communicate with family or friends
  7. Getting support from hospital doctors and nurses
  8. Able to return to work or usual home activities
  9. Feeling comfortable and in control
  10. Having a feeling of general well-being
  11. Moderate pain
  12. Severe pain
  13. Nausea or vomiting
  14. Feeling worried or anxious
  15. Feeling sad or depressed

SECONDARY OUTCOMES:
NRS score for rest and coughing pain | at 1, 6, 24, 48 hours after surgery
  Postoperative pain at rest and during coughing was assessed by NRS score with a range of 0 to 10 (0=no pain, 10=the worst possible pain)
consumption of opioid converted to IV morphine equivalents | during 24 hours after surgery
  opioids given postoperatively converted to IV morphine equivalents
the incidence of postoperative hypotension | during 48 hours after surgery
  Adverse reactions related to opioid
the incidence of nausea and vomiting | during 48 hours after surgery
  Adverse reactions related to opioid
the incidence of pruritus | during 48 hours after surgery
  Adverse reactions related to opioid
the incidence of respiratory depression | during 48 hours after surgery
  Adverse reactions related to opioid
time to urethral catheter removal in hours | through study completion, an average of 24-36 hours
  Time tourethral catheter removal after surgery
postoperative hospital stay in days | through study completion, an average of 5-7 days
  The time from operation to discharge
intra-operative opioid requirements | through the anesthesia process, an average of 1.5-2.5h
  opioids given intra-operatively
the block-related outcomes | through study completion, an average of 5-7 days
  the incidence of block-related complications (accidental intravascular injection, local anaesthetic systemic toxicity, haematoma and pneumothorax); and incidence of patient-reported transient neurological complications (paraesthesia or sensory deficit)
the Brief Pain Inventory | at 3 months after surgery.
  The Brief Pain Inventory instrument assesses 2 domains: pain and pain-related interference with physical and emotional functioning.
  1. pain at its worst in the last 24 hours
  2. pain at least in the last 24 hours
  3. describe your pain on average
  4. how much pain do you have right now
  5. interference with general activity
  6. interference with working ability
  7. interference with work
  8. interference with mood
  9. interference with relations with other people
  10. interference with sleep
  11. interference with enjoyment of life

CONTACTS AND LOCATIONS:
Overall Officials: Huifang Jiang, MD, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
Yes: There is a plan to make IPD and related data dictionaries available.
Supporting Information: Study Protocol, SAP
Time Frame: starting about 6 months after publication
Access Criteria: We will share data on ClinicalTrials.gov, and data sharing will be always available.

REFERENCES:
- [Derived] Gu B, Huang ZX, Zhou HD, Lian YH, He S, Ge M, Jiang HF. A Randomized Controlled Trial of Adding Deep Parasternal Intercostal Plane Block to Interpectoral-Pectoserratus Plane Block in Breast Cancer Surgery. Anesth Analg. 2025 May 1;140(5):1188-1194. doi: 10.1213/ANE.0000000000007218. PMID 39453840